CLINICAL TRIAL: NCT06430905
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Arenavirus-based Vector Therapy HB-502 and HB-501 in People With HIV on Suppressive Antiretroviral Treatment
Brief Title: Safety, Reactogenicity and Immunogenicity of HB-502 and HB-501 Versus Placebo in People With HIV on Suppressive ART
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision
Sponsor: Hookipa Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-500-001
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
Keywords: human immunodeficiency virus; HIV; vaccine; immunotherapy; arenavirus; genetic vector; antiretroviral therapy; ART
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HB-502 and HB-501 alternating 2-vector therapy (Dose Level 1) OR placebo (Experimental): Intramuscular injection of HB-502 and HB-501 alternating 2-vector therapy at Dose Level 1 OR placebo every 8 weeks for 24 weeks (injections at Weeks 0, 8, 16, and 24).
  Interventions: Biological: HB-502 and HB-501 alternating 2-vector therapy Dose Level 1; Other: Placebo
- HB-502 and HB-501 alternating 2-vector therapy (Dose Level 2) OR placebo (Experimental): Intramuscular injection of HB-502 and HB-501 alternating 2-vector therapy at Dose Level 2 OR placebo every 8 weeks for 24 weeks (injections at Weeks 0, 8, 16, and 24).
  Interventions: Biological: HB-502 and HB-501 alternating 2-vector therapy Dose Level 2; Other: Placebo

INTERVENTIONS:
Biological: HB-502 and HB-501 alternating 2-vector therapy Dose Level 1 — Administration of HB-502 and HB-501 alternating 2-vector therapy to 10 participants.
  Arms: HB-502 and HB-501 alternating 2-vector therapy (Dose Level 1) OR placebo
Biological: HB-502 and HB-501 alternating 2-vector therapy Dose Level 2 — Administration of HB-502 and HB-501 alternating 2-vector therapy to 10 participants.
  Arms: HB-502 and HB-501 alternating 2-vector therapy (Dose Level 2) OR placebo
Other: Placebo — Administration of placebo to 5 participants.

SUMMARY:
This is a study of HB-502 and HB-501 alternating 2-vector therapy in people living with human immunodeficiency virus (HIV) who are taking antiretroviral treatment (ART).

The benefits of available ART are short-lived and eventually there is a return of rapid HIV replication and higher viral copy number after a period of initial improvement of infection. The study treatment made of HB-502 and HB-501 is designed to train the body to recognize and fight parts from substances found in HIV.

This trial studies the safety, tolerability, and ability of HB-502 and HB-501 to stimulate an immune response against HIV in people living with HIV.

Participants will receive the study treatment by injection into the muscle every 8 weeks for a duration of 24 weeks, which is followed by another 24 weeks to continue looking closely at the safety profile and anti-HIV immune reaction after the last dose of study treatment.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1b, randomized, double-blind, placebo-controlled, multicenter study of HB-502 and HB-501 alternating 2-vector therapy in participants with HIV who are in overall good health and on suppressive ART. The study will evaluate the safety, reactogenicity, and immunogenicity of HB-502 and HB-501 alternating 2-vector therapy.

HB-502 and HB-501 are genetically engineered replicating vectors based on the arenaviruses Pichinde virus and lymphocytic choriomeningitis virus, respectively. The HB-502 and HB-501 vectors have been engineered to deliver HIV antigens derived from parts of key, immunogenic regions of HIV type 1 (HIV-1) proteins that are highly conserved within HIV-1 clade B variants. The designed immunogens differ from each other by their amino acid sequence allowing for coverage of >80% of circulating HIV-1 viral variants.

Two different dose levels (Dose Level 1 and Dose Level 2) of HB-502 and HB-501 alternating 2-vector therapy or placebo will be administered intramuscularly every 8 weeks for 24 weeks (i.e., 4 doses at Weeks 0, 8, 16, and 24), which is followed by a 24-week follow-up period.

In total, approximately 30 participants aged 18 to 65 years will be enrolled in this study to receive HB-502 and HB-501 alternating 2-vector therapy or placebo.

About 5 Investigators and study sites in the United States are expected to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 to 65 years of age.
* Confirmed HIV infection as documented by medical records or confirmatory HIV testing at screening.
* Must be on stable suppressive antiretroviral treatment (ART) for at least 48 weeks prior to screening.
* Must have plasma HIV RNA levels of <50 copies/mL (or lower limit of quantitation) for at least 48 weeks prior to enrollment.
* Must have a cluster of differentiation (CD)4+ cell count >450 cells/mm3 and CD4+ cell % of ≥15% obtained within 40 days prior to enrollment.
* Is in good general health according to the clinical judgment of the site Investigator.

Exclusion Criteria:

* History of hypersensitivity or other contraindication to any of the components of the study interventions as determined by the Investigator.
* HIV-associated malignancy according to the National Cancer Institute (including Kaposi's sarcoma), and any type of lymphoma or virus-associated cancers.
* History of HIV-associated neurocognitive disease or progressive multifocal leukoencephalopathy.
* More than stage 2 HIV-related illness based on the Revised Surveillance Case Definition for HIV Infection (CDC 2014).
* Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery within 156 weeks (i.e., 3 years) prior to enrollment.
* Known history of hepatitis B virus (defined as hepatitis B surface antigen reactive) or known active hepatitis C virus infection (defined as hepatitis C virus RNA is detected [qualitative]).
* Current untreated or incompletely treated active TB disease or untreated latent TB infection.
* Has any serious or uncontrolled medical disorder that, in the opinion of the Investigator, may increase the risk associated with study participation or study treatment administration, impair the ability of the participant to receive study treatment, or interfere with the interpretation of the study results.
* Is a previous or current recipient of an investigational HIV vaccine (previous placebo/control recipients are not excluded).
* Received non-HIV experimental vaccine(s) within the last 1 year.
* Has congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site Investigator, such as history of systemic corticosteroids (long-term use), immunosuppressive anti-cancer or other immunosuppressive agents, interleukins, systemic interferons, systemic chemotherapy, or other medications considered significant by the Investigator within 24 weeks prior to the start of study therapy.
* Received blood products or immunoglobulin within 16 weeks prior to enrollment.
* Received systemic steroids at a dose of ≥10 mg/day (prednisone equivalent) for <30 within 14 days or for ≥30 days within 28 days of first dose of study treatment.
* Received any vaccine within 4 weeks prior to enrollment.
* Initiated antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary).
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or contraindicate participation in this study, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
* Is pregnant or breastfeeding or expecting to conceive or father children starting with the screening visit through a minimum of 12 weeks after the last dose of trial treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From first dosing until 48 weeks after first dosing
  Assess the safety of HB-502 and HB-501 alternating 2-vector therapy compared with placebo by monitoring the type, frequency, and severity of unsolicited treatment-emergent and serious AEs, using the Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric AEs, Corrected Version 2.1, July 2017.
Number of participants with local injection site reactions | From first dosing until 48 weeks after first dosing
  Assess the frequency and type of solicited local injection site reactions in response to HB-502 and HB-501 alternating 2-vector therapy compared with placebo, using the DAIDS Table for Grading the Severity of Adult and Pediatric AEs, Corrected Version 2.1, July 2017.
Number of participants with systemic reactogenicity events | From first dosing until 48 weeks after first dosing
  Assess the frequency and type of solicited systemic reactogenicity events in response to HB-502 and HB-501 alternating 2-vector therapy compared with placebo, using the DAIDS Table for Grading the Severity of Adult and Pediatric AEs, Corrected Version 2.1, July 2017.

SECONDARY OUTCOMES:
Determine the magnitude of the cellular immune response against HIV-1 induced by HB-502 and HB-501 alternating 2-vector therapy compared with placebo | From first dosing until 48 weeks after first dosing
  Assess changes from baseline in the magnitude of T cell response specific to the transgenes harbored in HB-502 and HB-501.
Determine the breadth of the cellular immune response against HIV-1 induced by HB-502 and HB-501 alternating 2-vector therapy compared with placebo | From first dosing until 48 weeks after first dosing
  Assess changes from baseline in the breadth of T cell responses to the different transgenes harbored in HB-502 and HB-501.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Development, Study Director — Hookipa Biotech GmbH
Locations (5):
- United States (5):
  - Orlando Immunology Center (OIC), Orlando, Florida
  - The Hope Clinic at Emory University, Decatur, Georgia
  - Brigham and Women´s Hospital, Boston, Massachusetts
  - Beth Israel Deaconness Medical Center (BIDMC), Boston, Massachusetts
  - Perelman Center for Advanced Medicine at the Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania